CLINICAL TRIAL: NCT01458496
Title: Health Coaching to Effect Lifestyle Behaviour Change: A Randomized Trial of Individuals With Pre-disease
Brief Title: Health Coaching to Effect Lifestyle Behaviour Change
Acronym: HC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marshal Godwin (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Marshal Godwin, Professor, Faculty of Medicine, Memorial University of Newfoundland
Organization: Memorial University of Newfoundland (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 243401
Record Dates: First submitted 2011-10-18; First posted 2011-10-24 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Prediabetes; Prehypertension
MeSH Terms: conditions — Prediabetic State; Prehypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health Coaching (Experimental)
  Interventions: Behavioral: Health Coaching
- Usual Care -Control (No Intervention): Patients assigned to the control (usual care) group will be advised to seek standard lifestyle counselling from their primary care physician.

INTERVENTIONS:
Behavioral: Health Coaching — The intervention will take approximately six months to complete. A combination of group and individual face-to-face meetings will be used. Participants will be divided into groups of 20 for group meetings. Groups will be brought together for a group coaching session at the beginning and the end of the coaching process (i.e., intervention). Each participant will also receive four individual coaching sessions with the health coach and will be able to avail of three one-hour telephone coaching sessions during the six month intervention. Participants will be encouraged to utilize telephone coaching for key support periods.
  Arms: Health Coaching

SUMMARY:
A health coaching intervention in those with pre-disease (pre-hypertension or pre-diabetes) but without pre-existing cardiovascular disease will effectively help participants change their lifestyle behaviour and prevent or delay onset of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-60 years
* Last recorded fasting blood glucose between 6.0 abd 6.9 mmol/L
* Last recorded blood pressure between 130-139 mmHG systolic and/or85-89 mmHG diastolic

Exclusion Criteria:

* Diagnosis of diabetes on the chart
* Diagnosis of hypertension on the chart
* taking an anti-diabetic medication
* taking an antihypertensive medication

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 219 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in lifestyle behaviours as measured by the Simple Lifestyle Indicator Questionnaire | baseline, 6 months, 12 months

SECONDARY OUTCOMES:
Change from baseline in Self-efficacy | baseline, 6 months, 12 months
Change from baseline in score on the Framingham-based Global Risk Assessment | baseline, 6 months, 12 months
Change from baseline in blood pressure as measured by the BpTRU device | baseline, 6 months, 12 months
Change from baseline in fasting blood glucose and HbA1c as measured by the Cholestech Analyser | baseline, 6 months, 12 months
Change from baseline in health related quality of life | baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Godwin, MD, MSc, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada